CLINICAL TRIAL: NCT07345897
Title: Advancing Cervical Cancer Screening Through Emergency Department-based Self-Sampling
Brief Title: Emergency Department-based Cervical Cancer Screening Through Self-sampling
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Beau Abar, Professor, University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 00011046
Record Dates: First submitted 2026-01-07; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: HPV; HPV Associated Cancers; HPV Cancers; Cervical Cancer Screening; Cervical Cancer (Early Detection)
Keywords: HPV Screening; Cervical cancer screening; HPV; Cervical cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Arm (Experimental): Participants will be provided the opportunity to self- sample for HPV during their ED visit. Participants will be (1) briefly instructed by study staff on how to self-sample using a defined instructional script written at an elementary reading level, (2) provided with a packaged swab, and (3) invited to self- sample privately in their ED room or in one of the private ED restrooms. Once self sampling has been completed, the study staff will then transfer the swab to a vial of transport media and forward the specimens to the laboratory for analysis. Participants recruited to the intervention arm that subsequently decline to or are unable to self-sample in the ED will remain in the study and will receive referral for clinic-based screening.
  Interventions: Diagnostic Test: Cervical Cancer Screening

INTERVENTIONS:
Diagnostic Test: Cervical Cancer Screening — Subjects will perform self sampling for cervical cancer.

SUMMARY:
This project will compare the uptake of cervical cancer screening through ED HPV sampling among patients presenting to the ED.

DETAILED DESCRIPTION:
This is a single-arm pilot trial with a prospectively enrolled sample. The participants who complete the screening survey and are determined to be adherent (n ~ 600) will be notified that they appear to be adherent with current screening guidelines, and their participation ends at this point. These participants will be considered screen failures for study purposes. Women and transgender/non-binary individuals with a cervix, aged 30-65, will be recruited from a high-volume urban ED. Follow-up will occur at 150 days to determine CC screening activity, perceived and concrete barriers to care, and participant experiences with the intervention. Electronic Health Record (EHR) review will be conducted to corroborate participants' reports of screening activities and assess completion of clinic-based testing and clinical endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Cisgender women and transgender/non-binary individuals with a cervix,
* Age 30 - 65 years, and demonstrating decisional capacity to consent to participate with no known exclusion criteria present.

Exclusion Criteria:

* Past hysterectomy with cervical removal
* Known infection with HIV (as screening recommendations for people with HIV differ from the general population)
* Inability to consent (e.g., lacking decisional capacity, intoxicated, or in distress)
* Current pregnancy or in the three months after giving birth
* Use of vaginal ovules, creams or washes, vaginal contraceptives or condoms within past 3 days
* Sexual intercourse or transvaginal ultrasound scans or gynecological examinations within past 2 days

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Uptake of cervical cancer screening from self-sampling in the ED | In about 150 days of enrollment
  Number of subjects referred for additional screening who follow through with next steps in the screening process.

IPD SHARING:
Plan to Share IPD: Undecided
No decision has been made to share individual participant data however there is no current plan to share on an individual basis.